CLINICAL TRIAL: NCT00180206
Title: Prospective, Non-Randomised, Non-Comparative Multicentric Investigation of the Functional and Radiological Result and Subjective Patient Outcome After Implantation of a Hip Resurfacing Endoprosthesis (Birmingham Hip Resurfacing)
Brief Title: Birmingham Hip Resurfacing (BHR) Study: Implantation of a Hip Resurfacing Endoprosthesis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DresdenU
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-01-16 (Estimated); Status verified 2005-09

CONDITIONS: Arthritis
Keywords: Arthritis; Hip; Hip arthroplasty; Hip resurfacing arthroplasty
MeSH Terms: conditions — Arthritis

INTERVENTIONS:
Device: Birmingham Hip Resurfacing

SUMMARY:
The purpose of this study is the investigation of the functional and radiological results and subjective patient outcome after the implantation of a hip resurfacing endoprosthesis (Birmingham hip resurfacing).

DETAILED DESCRIPTION:
High volumetric wear of polyethylene was the main factor in periprosthetic bone resorption and failure of historic hip resurfacing prosthesis. Metal-on-metal devices reduce the wear substantially and may solve this problem. The purpose of this study is the investigation of the functional and radiological result and subjective patient outcome after implantation of a hip resurfacing endoprosthesis (Birmingham Hip Resurfacing) during the first two years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological signs of coxarthritis
* Implantation of a total hip replacement indicated
* Informed consent

Exclusion Criteria:

* Osteoporosis
* Tumor
* Acute infection
* Higher grade congenital dysplasia of the hip
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-01; Study Completion 2008-12

PRIMARY OUTCOMES:
Functional result
Radiological result
Subjective patient outcome

SECONDARY OUTCOMES:
Perioperative and postoperative complication rate
Revision rate

CONTACTS AND LOCATIONS:
Overall Officials: Klaus-Peter Guenther, Prof., Principal Investigator — Department of Orthopaedic Surgery, University Hospital Carl Gustav Carus, Technical University of Dresden
Locations (1):
- Department of Orthopaedic Surgery, University Hospital, Technical University of Dresden, Dresden, Germany